CLINICAL TRIAL: NCT06036303
Title: Nasr Fascial Closure: A Novel Device for Fascial Closure in Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ClinAmygate (Other)
Collaborators: Aswan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR00C1945
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cholecystolithiasis
Keywords: Laparoscopic removal
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasr Fascial Closure Device (Experimental)
  Interventions: Device: Nasr fascial closure device
- Berci Fascial Closure Device (Active Comparator)
  Interventions: Device: Berci Fascial Closure Device

INTERVENTIONS:
Device: Nasr fascial closure device — Nasr fascial closure device is a novel device for fascial closure
  Arms: Nasr Fascial Closure Device
Device: Berci Fascial Closure Device — Berci Fascial Closure Device is a known device for fascial closure
  Arms: Berci Fascial Closure Device

SUMMARY:
The study will investigate the efficacy and safety of a new fascial closure device "Nasr Fascial Closure Device" compared to the Karl Storz Berci Fascial Closure Device 26173AM.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* eligible for Laparoscopic cholecystectomy

Exclusion Criteria:

* refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
duration of port site closure | 1 day
  Duration in seconds
Rate of failure of port site | 1 day
  Rate of failure to close the port site

SECONDARY OUTCOMES:
Incidence of port site infection | 1 month
  Incidence of infection of the port site
Incidence of port site hernia | 6 weeks
  Incidence of hernia at the port site

CONTACTS AND LOCATIONS:
Overall Officials: Mohie El-Din M Madany, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt